CLINICAL TRIAL: NCT05271461
Title: Effect of Low Level Laser Therapy on Hyper Coagulability in Patients With Covid-19
Brief Title: COVID-19 Hyper Coagulability Care by LLLT
Acronym: LLLT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Enas Wagdy Elsaid Ahmed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: COVID-19 LLLT.
Record Dates: First submitted 2022-02-14; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Two groups of 30 patients, 1st circulatory exercise, 2nd LLLT and circulatory exercises.
Who Masked: Care Provider
Masking Description: circulatory exercise only, circulatory exercises and LLLT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Circulatory exercises group . (Active Comparator): Circulatory exercises.
  Interventions: Other: Circulatory exercises
- LLLT group . (Experimental): Low level laser Therapy + circulatory exercises.
  Interventions: Radiation: Low level laser Therapy; Other: Circulatory exercises

INTERVENTIONS:
Radiation: Low level laser Therapy — Pin pointed application of low level laser on 15 acupuncture points each point 1 min time of application 15 min.
  Arms: LLLT group .
Other: Circulatory exercises — Active assisted or against mild resistance. Supine with leg up position 18degrees measured by the bed water balance in side rails.
  If patient is not comfortable according to the modified Borg scale or contra indicated for the position then assume the supine position.
  The subject will have A 3 min rest period to acclimatize themselves to each position.
  The ankle pumping exercises consisted of simple repetitions of dorsiflexion 1 sec and planter- flexion for 1 sec with three different exercise intervals:
  * repeated dorsiflexion and planter-flexion with no rest (no rest exercise).
  * repeated dorsiflexion and planter-flexion with a 2 sec rest period (2 sec rest exercise).
  * repeated dorsiflexion and planter-flexion with 4sec rest period (4sec rest exercise).
  Subjects will have practiced ankle pumps before the exercise to get familiar and be educated about the procedure.

SUMMARY:
COVID-19 clotting Safety

DETAILED DESCRIPTION:
Covid-19 patients have liability for hyper coagulability, low level laser Therapy improve circulation and decrease liability for hyper coagulability accompanied with circulatory exercises .

ELIGIBILITY:
Inclusion Criteria:

* BMI from 18.5 to 29.9 kg/m2
* Moderate elevated percentage of coagulative factors for COVID-19 Diagnosis:
* Nasopharyngeal swab
* Sepsis induced coagulopathy score>4
* D_dimer≥0,5mg/L
* Fibrinogen>2,5gm/L
* C_reactive protein≥10mg/L
* Lymphocyte count<1,500mm3
* Platelet count<150,000mm3
* Prothrombin time increase>3sec
* Activated partial thromboplastin time increase>5sec
* Same level of physical activity
* Patients can swallow tablets
* CT scan screening method for COVID-19 Diagnosis
* Physical examination

Exclusion Criteria:

* hyper tension
* Cognitive impairment e.g (delirium)
* Diabetes mellitus both types dependant or non
* Disabled musculoskeletal Disorders e.g hemi paresis
* Coronary artery diseases and heart failure
* DVT
* Stroke, bone disease, renal failure, pulmonary embolism
* Vitamins deficiency
* 6 months post large surgeries
* Alcohol intake and smokers
* Thyroid diseases

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-04 (Estimated); Study Completion 2022-06-04 (Estimated)

PRIMARY OUTCOMES:
Circulatory group laboratory investigation. | Monthly (an average of two months)
  D-dimer≥.5mg/dL, fibrinogen>2.5mg/dL
  To examine COVID-19 recovery.
Circulatory group: CBC analysis. | Daily (an average of two months)
  Lymphocyte count<1.500mm3, Platelet count<150.000mm3, to examine COVID-19 recovery.
Circulatory group (PT, PTT). | Bi weekly (an average of two months)
  Prothrombin time>3 sec, activated partial thromboplastin time>5 sec to examine COVID-19 recovery.
Circulatory group physical examination. | Every two days (an average of two months)
  by visual analog scale is horizontal line 100mm length the ends defined as extreme limit of the parameter measured (symptom, pain, health) orientated from the left (the worst) the right (the best) 3 times per week to detect DVT.
Circulatory group. BMI. | Day one
  weight kg on height m2 to detect liability for DVT.
Especially Lab investigation. | Baseline
  C-reactive protein ≥10mg/l for diagnosis of the recovery.

SECONDARY OUTCOMES:
LLLT group laboratory investigation. | Monthly (an average of two months)
  D-dimer≥,5mg/dl, fibrinogen>2.5mg/dl, c-reactive protein≥10mg/dl to examine COVID-19 recovery.
  Fibrinogen
LLLT group CBC analysis. | Daily (an average of two months)
  lymphocyte count<1,500mm3, platelet count<150,000mm3, for examine COVID-19 recovery.
LLLT group. {PTT, PT}. | Bi weekly (an average of two months)
  Prothrombin time>3 sec, activated partial thromboplastin time>5sec to examine COVID-19 recovery.
LLLT group physical examination. | Every two days (an average of two months)
  by visual analog scale is a straight horizontal line of fixed length 100mm the end is extreme limit of the parameter measured (symptom, pain, health) orientated from the left (the worst) to the right (the best) 3times per week to detect DVT.
LLLT group. BMI. | Day one
  Weight kg/height m2 to detect liability for DVT.
Specifically Lab investigation. | Baseline
  C_reactive protein≥10mg/l.help diagnosis of the recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Enas Dr Ahmed, BSC, Principal Investigator — Physical therapy faculty CairoU.
Locations (1):
- Physical therapy faculty, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agaiby AD, Ghali LR, Wilson R, Dyson M. Laser modulation of angiogenic factor production by T-lymphocytes. Lasers Surg Med. 2000;26(4):357-63. doi: 10.1002/(sici)1096-9101(2000)26:43.0.co;2-o. PMID 10805940
- [Background] Emami A, Javanmardi F, Pirbonyeh N, Akbari A. Prevalence of Underlying Diseases in Hospitalized Patients with COVID-19: a Systematic Review and Meta-Analysis. Arch Acad Emerg Med. 2020 Mar 24;8(1):e35. eCollection 2020. PMID 32232218
- [Background] ConnorsJ.M.,LevyJ.H(2020).Thromboinflammation and the hyper coagulability of COVID-19.JThromb Haemost https://doi.org/10.1111/jth.14849.